CLINICAL TRIAL: NCT01646424
Title: Validation of Questionnaire and Assessment of Patient Satisfaction for Budesonide/Formoterol Fix Combination DPI in COPD
Brief Title: Validation of Questionnaire and Assessment of Patient Satisfaction for Budesonide/Formoterol Fix Combination Dry Powder Inhalers (DPI) in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RTR-XXX-2012/1
Record Dates: First submitted 2012-07-19; First posted 2012-07-20 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD,; Patient satisfaction,; fix combination,; NIS Turkey,; turbuhaler,; FSI-10
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to describe patient preferences on budesonide/formoterol fix dose combination for the treatment of their COPD, and to find those factors more strongly associated to a better attitude to medication.

DETAILED DESCRIPTION:
Validation of questionnaire and assessment of patient satisfaction for budesonide/formoterol fix combination DPI in COPD

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent and to be an outpatient
* Clinical diagnosis of COPD according to ICD-10 classification, females and males, aged ≥ 40 years
* To be prescribed a fixed dose combination of inhaled budesonide/formoterol fix combination at least 3 months before the study start

Exclusion Criteria:

* Pregnancy for women
* Use of inhaled medication via a metered dose inhaler (pMDI)
* Currently participating in randomized clinical trials and being included in this study once

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes ≥ 40 years of age, diagnosed with COPD (according to ICD-10 criteria) and receiving budesonide/formoterol fix dose combination treatment by means of inhaler devices. The first prescription must be given at least 3 months prior to the study start and patient inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Feeling of Satisfaction with Inhaler (FSI-10) Questionnaire in COPD Turkish population. | During 1 month, up to September 2012
  The FSI-10 is a self-completed 10-item questionnaire to assess patient opinions regarding ease or difficulty of use, portability, and usability of devices for delivery of inhaled medications. Each of the 10 items has 5 response options from poorer to greater ease of use, scored 1 to 5, respectively. The minimum score is 10 whereas the maximum is 50.

SECONDARY OUTCOMES:
Socio-demographics profile | During 1 month, up to September 2012
  Socio-demographics parameters: Age; Gender; Educational level; Place of residence (urban / rural); Living alone or accompanied.
Clinical characteristics | During 1 month, up to September 2012
  Clinical characteristics parameters:Current disease grade; Date of COPD diagnosis
Treatment-related information | During 1 month, up to September 2012
  Date of first prescription for Turbuhaler; Concomitant treatments for COPD
Inhaler use | During 1 month, up to September 2012
  Specifically for evaluating real-life patterns of use and usage knowledge of the dry-powder inhaler (Turbuhaler) that delivers budesonide / formoterol fix combination, a specific checklist of the key features of the inhalation technique.Preference with the inhaler she/he is using will be assessed based on patient reported outcomes.
Site characteristics | During 1 month, up to September 2012
  Type of the hospital: state, university, private

CONTACTS AND LOCATIONS:
Overall Officials: Mujgan Ates, DR, Study Director — AZ MC Turkey; Akin Kaya, PROF.DR., Principal Investigator — Ankara University Faculty of Medicine, Chest Diseases Department
Locations (20):
- Turkey (Türkiye) (20):
  - Research Site, Adana
  - Research Site, Afyonkarahisar
  - Research Site, Ankara
  - Research Site, Ayd?n
  - Research Site, Balıkesir
  - Research Site, Bartın
  - Research Site, Çankırı
  - Research Site, Elâzığ
  - Research Site, Gaziantep
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kayseri
  - Research Site, Kocaeli
  - Research Site, Konya
  - Research Site, Manisa
  - Research Site, Mersin
  - Research Site, Rize
  - Research Site, Sakarya
  - Research Site, Samsun
  - Research Site, Yozgat